CLINICAL TRIAL: NCT03238300
Title: Neuroscience-Informed Treatment Development for Adolescent Alcohol Use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Lindsay Squeglia, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00058771; K23AA025399 (NIH)
Record Dates: First submitted 2017-07-31; First posted 2017-08-03 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Alcohol Drinking; Control
Keywords: adolescent
MeSH Terms: conditions — Alcohol Drinking | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- N-Acetylcysteine, then Placebo (Experimental): Participants first received N-Acetylcysteine 600mg capsules by mouth, two pills twice daily will be taken for 10 days. After washout for 11 days, they then received placebo capsules mimicking N-Acetylcysteine (two pills, twice daily) will be taken for 10 days.
  Interventions: Drug: N-Acetylcysteine; Drug: Placebo Oral Capsule
- Placebo, then N-Acetylcysteine (Experimental): Participants first received placebo capsules mimicking N-Acetylcysteine (two pills, twice daily) will be taken for 10 days. After washout for 11 days, they then received N-Acetylcysteine 600mg capsules by mouth, two pills twice daily will be taken for 10 days.
  Interventions: Drug: N-Acetylcysteine; Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: N-Acetylcysteine — N-Acetylcysteine; 600mg capsules by mouth, two pills twice daily (total 2400 mg/day). Participants will undergo MRI (including magnetic resonance imaging and functional MRI during an alcohol cue reactivity task) at baseline, after 10 days of N-Acetylcysteine and after 10 days of placebo.
Drug: Placebo Oral Capsule — N-acetylcysteine-matched placebo tablet two pills twice daily. Participants will undergo MRI (including magnetic resonance imaging and functional MRI during an alcohol cue reactivity task) at baseline, after 10 days of N-Acetylcysteine and after 10 days of placebo.

SUMMARY:
This study will examine the effect of N-Acetylcysteine (NAC), an over-the-counter antioxidant supplement, on brains of youth (ages 15-19) using magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
55 adolescents will receive, in a counterbalanced order, a 10-day course of NAC 1200 mg twice daily and a subsequent 10-day course of matched placebo twice daily, separated by 11 days. Urine and blood samples will be collected at baseline and urine samples again before and after each course of medication treatment. Participants will receive a 1- hour MRI scan at baseline and after each treatment trial.

ELIGIBILITY:
Inclusion criteria: Participants were between the ages of 15-19 and may or may not have used alcohol. All participants in the alcohol-using group met criteria for heavy drinking, based on quantity and frequency of drinking (Squeglia et al. 2011; Squeglia et al. 2012) (see Figure 2).

Exclusionary criteria: Not having a parent to consent (for those under age 18); history of alcohol treatment or treatment-seeking; current DSM-5 diagnosis of moderate or severe substance use disorder other than alcohol or cannabis (American Psychiatric Association 2013); positive urine toxicology screen for narcotics, amphetamines, sedatives, hypnotics, or opiates (not prescribed by a doctor); alcohol withdrawal (> 10 on the Clinical Institute Withdrawal Assessment for Alcohol (Sullivan et al. 1989); medical conditions or medications that contraindicate taking NAC; current use of N-acetylcysteine or any supplement containing N-acetylcysteine (must agree not to take any such supplement throughout study participation); medical history of severe asthma (uncontrolled with medication); history of a serious medical, psychiatric, or neurological problem that could affect neural response, brain development, or study participation, including diabetes, seizure disorder, and severe head injury with loss of consciousness; history of learning disability, pervasive developmental disorder, or other condition requiring special education; current use of psychoactive medications that affect cerebral blood flow; non-correctable visual or hearing problems; non-fluent in English; MRI contraindications (e.g., braces, claustrophobia, irremovable metal implants or piercings); (for females) pregnancy or refusal to use reliable methods of birth control; refusal of blood draw, abstinence from alcohol for >14 days before participation, and use of alcohol <12 hours before scanning (confirmed with breathalyzer). While cigarette and marijuana use will not be exclusionary, we will exclude any participants who are daily users of cannabis or tobacco.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay M Squeglia, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 57 participants were screened for eligibility between October 16, 2017 and February 18, 2022 at the Medical University of South Carolina.
Pre-assignment Details: 35 of 57 were randomized. Of those not randomized, 12 were ineligible, 6 declined to participate, and 4 withdrew or were withdrawn during the baseline visit.
Groups:
- N-Acetylcysteine, Then Placebo: N-Acetylcysteine 600mg capsules by mouth, two pills twice daily will be taken for 10 days. After washout for 11 days, placebo capsules mimicking N-Acetylcysteine (two pills, twice daily) will be taken for 10 days.
- Placebo, Then N-Acetylcysteine: Placebo capsules mimicking N-Acetylcysteine (two pills, twice daily) will be taken for 10 days. After washout for 11 days, N-Acetylcysteine 600mg capsules by mouth, two pills twice daily will be taken for 10 days
Period: Baseline (Before Intervention)
Arm/Group | N-Acetylcysteine, Then Placebo | Placebo, Then N-Acetylcysteine
Started | 18 | 17
Completed | 18 | 16
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: First Intervention (10-Days)
Arm/Group | N-Acetylcysteine, Then Placebo | Placebo, Then N-Acetylcysteine
Started | 18 | 16
Completed | 18 | 16
Not Completed | 0 | 0
Period: Washout Period (11-Days)
Arm/Group | N-Acetylcysteine, Then Placebo | Placebo, Then N-Acetylcysteine
Started | 18 | 16
Completed | 17 | 16
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention (10-Days)
Arm/Group | N-Acetylcysteine, Then Placebo | Placebo, Then N-Acetylcysteine
Started | 17 | 16
Completed | 15 | 16
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-Acetylcysteine, Then Placebo | Placebo, Then N-Acetylcysteine | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 18.90 (0.75) | 18.79 (0.60) | 18.85 (0.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 9 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 15 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Quantifying the Difference in Glutamate Levels (mmol/kg) During N-Acetylcysteine Versus Placebo in the Anterior Cingulate Brain Region.
Description: Using magnetic resonance spectroscopy and a within-subjects design, we will determine the effect of N-Acetylcysteine versus placebo on modulating anterior cingulate glutamate levels in adolescents. Values provided are absolute values (mmol/kg) at the end of each intervention period. Due to complexities of this method, "normal" levels of glutamate are not known; thus, we cannot make conclusions about the meaning of "higher" or "lower" glutamate levels when comparing N-acetylcysteine to placebo.
Time Frame: 31 days total (levels compared after 10 days on N-Acetylcysteine and 10-days of placebo with 11 day washout period in between)
Measure: Mean (Standard Deviation); unit: mmol/kg
Groups:
- N-Acetylcysteine: N-Acetylcysteine 600mg capsules by mouth, two pills twice daily will be taken for 10 days
- Placebo: Placebo capsules mimicking N-Acetylcysteine (two pills, twice daily) will be taken for 10 days
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 31 | 31
mmol/kg | 15.7527667 (0.748460934) | 15.6265229 (0.778392692)
Statistical Analysis 1: Comparison: N-Acetylcysteine vs Placebo; With 31 participants, the study has 99% power to detect such effects on glutamate levels (calculated based on d =1.13 [reported in Schmaal et al., 2012], α = 0.05, two-tailed). We used linear mixed effects models with random intercepts with medication, visit, and sequence. Baseline metabolite levels and brain tissue composition [GM:BM = GM/(GM+WM)], cannabis use (days), and alcohol use disorder status (Yes/No) were included as covariates; Test type: Superiority; p > 0.05, Mixed Models Analysis — P-value >0.05 for main effect of medication (N-acetylcysteine vs. placebo); Random intercepts were used; partial eta squared = 0.02, 95% CI 2-sided [0.00 to 0.22]

2. Primary Outcome: Change in Neural Reactivity (as Measured by BOLD: Blood Oxygen Level-Dependent Response) in Reward Regions During Alcohol-cue Reactivity Task.
Description: Assessing the change in neural reactivity to alcohol cues after each round of medication: Placebo vs. N-Acetylcysteine.
  Cue reactivity is a type of learned response which is observed in individuals who use substances (e.g., alcohol) and involves significant physiological reactions to presentations of substance-related stimuli (i.e., alcohol images) in comparison to neutral images (e.g., non-alcoholic beverages ) measured by BOLD (Blood Oxygen Level-Dependent response). ROIs were (left and right hemisphere): amygdala, caudate, insula, nucleus accumbens, and putamen.
  Change in BOLD signal are reported in Z-scores. A Z-score of 0 would indicate there is no statistical difference in BOLD signal between alcohol images and non-alcohol beverage images. A higher Z-score would indicated a higher BOLD signal during alcohol images compared to non-alcohol beverage images. A lower Z-score would indicate a lower BOLD signal during alcohol images compared to non-alcohol beverage images.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- N-Acetylcysteine: N-Acetylcysteine 600mg capsules by mouth, two pills twice daily for 10 days.
  N-Acetylcysteine: N-Acetylcysteine pill.
- Placebo Oral Capsule: Placebo capsules by mouth, two pills twice daily for 10 days.
  Placebo Oral Capsule: Sugar pill to mimic.
Arm/Group | N-Acetylcysteine | Placebo Oral Capsule
Number analyzed (Participants) | 31 | 31
Z-score
  Left Amygdala | 0.649576194 (0.968974541) | 0.3018234193548 (0.841575583)
  Right Amygdala | 0.56294871 (0.999382512) | 0.210653871 (0.946731462)
  Left Caudate | 0.137316806 (0.970053483) | 0.110683871 (0.826040069)
  Right Caudate | 0.065642839 (1.100274051) | 0.031422161 (0.79443319)
  Left Insula | -0.258198161 (1.142477966) | 0.058738871 (0.846769387)
  Right Insula | -0.429143032 (1.2071406050607) | -0.169528194 (1.075103119)
  Left Nucleus Accumbens | 0.347468645 (1.0725798) | 0.2095879354838 (0.697815244)
  Right Nucleus Accumbens | 0.240204258 (1.151021574) | 0.072915871 (0.9231385308441)
  Left Putamen | -0.138118065 (0.894080737) | 0.225092871 (0.989678164)
  Right Putamen | -0.165481516 (0.818905961) | 0.058414516 (0.9453397543003)
Statistical Analysis 1: Comparison: N-Acetylcysteine vs Placebo Oral Capsule; Contrast of interest was alcohol beverages vs. non-alcohol beverages. We used linear mixed effects models with random intercepts with medication, visit, and sequence. Baseline reactivity levels for each ROI, cannabis use (days), and an alcohol use covariate (quantity, frequency, AUD status, or AUD severity - depending on which best fit the model) were included as covariates. ROIs included were (left and right hemisphere): amygdala, caudate, insula, putamen, and nucleus accumbens; Test type: Superiority; p > 0.05, Mixed Models Analysis — P-value >0.05 for main effect of medication (N-acetylcysteine vs. placebo) for all ROIs; Random intercepts were used for all models

ADVERSE EVENTS:
Time Frame: 31 days (10 days of first intervention, 11-day wash out, 10 days of second intervention) Intervention = N-acetylcysteine, then Placebo OR Placebo, then N-acetylcysteine
Description: Participants were asked about adverse events at every visit, either from a research assistant, principal investigator, medical clinician, or other study staff.
Groups:
- Washout Period: 11-days with no medication, but check in with study staff and assessment of AEs
- Baseline: Prior to first intervention
Arm/Group | N-Acetylcysteine | Placebo Oral Capsule | Washout Period | Baseline
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34 | 0/33 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/33 | 0/35
Other Adverse Events (participants affected / at risk) | 10/34 | 5/34 | 1/33 | 2/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetylcysteine (N=34) | Placebo Oral Capsule (N=34) | Washout Period (N=33) | Baseline (N=35)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Mild, causality: remote, no action taken
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) — Mild, Definitely Not Related, No Action Taken
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Mild, remotely related, no action taken
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Milld, Definitely not related, Referred to/seen by PCP
Skin and subcutaneous tissue disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mild, remotely related, no action taken
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) — Mild or moderate, possibly related, no action taken
Stomachache (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) — Mild, Possibly related, No action taken
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mild, Definitely not related, no action taken
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Moderate, definitely not related, Referred to/seen by PCP
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Mild, probably related, no action taken
Viral Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Mild, definitely not related, no action taken

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Detailed Protocol & General Statistical Analysis Plan (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT03238300/Prot_SAP_003.pdf
  • Statistical Analysis Plan: Detailed SAP (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT03238300/SAP_004.pdf
  • Informed Consent Form (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT03238300/ICF_005.pdf